CLINICAL TRIAL: NCT04945499
Title: The Evaluation of D-glucose Weighted Chemical Exchange Saturation Transfer (gluceoCEST)-Based Dynamic Glucose Enhanced(DGE) Magnetic Resonance Imaging（MRI） in Brain Tumor
Brief Title: The Application of Glucose CEST MR Imaging in Brain Tumor
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DGE CEST MR and brain tumor
Record Dates: First submitted 2021-03-23; First posted 2021-06-30 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Magnetic Resonance Imaging
Keywords: dynamic glucose enhanced; human brain tumor; chemical exchange saturation transfer
MeSH Terms: interventions — Glucose

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- D-glucose (Other): During the dynamic glucose scan, a brief hyperglycemic state was established by intravenous infusion of hospital-grade D50 glucose (D50, 25 g of dextrose in 50 mL of water sterile solution), followed by 20 mL of saline solution in 1 arm. The glucose infusion was performed using a power injector at an infusion rate of 0.2 mL/s, corresponding to total infusion times 250 seconds.
  Interventions: Drug: d-glucose

INTERVENTIONS:
Drug: d-glucose — using d-glucose as an contrast agent on CEST MR Imaging
  Other Names: 50% dextrose injection

SUMMARY:
Recently, natural D-glucose was suggested as a potential biodegradable contrast agent. The feasibility of using D-glucose for dynamic perfusion imaging was explored to detect malignant brain tumors based on blood brain barrier breakdown. Our study try to evaluate the feasibility of dynamic glucose enhanced(DGE) magnetic resonance imaging（MRI）in brain tumor, which based on D-glucose weighted chemical exchange saturation transfer (gluceoCEST).

DETAILED DESCRIPTION:
methods： Brain tumor patients were recruited. Time-resolved glucose signal changes were detected using chemical exchange saturation transfer (glucoCEST) MRI. Dynamic glucose enhanced (DGE) MRI was used to measure tissue response to an intravenous bolus of D-glucose. During the dynamic glucose scan, a brief hyperglycemic state was established by intravenous infusion of hospital-grade D50 glucose (D50, 25 g of dextrose in 50 mL of water sterile solution), followed by 20 mL of saline solution in 1 arm. The glucose infusion was performed using a power injector at an infusion rate of 0.2 mL/s, corresponding to total infusion times of 250 seconds. Performing contrast enhancement based on Gd-DTPA in 30 minutes later, which was used for comparison as golden standard.

The area of hyperintensity will be measured, which represents the area of brain tumor.

Differential test and Consistency analysis were used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a brain mass consistent with a primary brain tumor or metastatic brain tumor
* able to give consent and willingness to participate in this study.

Exclusion Criteria:

* presence of any ferromagnetic implant (cardiac pacemakers, aneurysm clip, etc.)
* pregnancy
* claustrophobia or anxiety disorder
* history of vertigo
* persons with diabetes mellitus (self-report or HbA1C >= 6.5%)
* Sickle cell disease
* persons taking prescription medicine for hypertension
* blood iron deficiency (Hb concentration < 11 g/dL or Hct < 32%)
* If volunteering for MRI: history of kidney disease and/or eGFR < 60.
* Middle-ear disorder
* double vision
* Seizure disorder
* Multiple myeloma
* Solid organ transplant
* History of severe hepatic disease/liver transplant/pending liver transplant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
CEST value of tumor lesion including tumor core/ necrosis/ cysis/ edema | 1 week
  the CEST value of tumor core and necrosis might higher than white matter

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2019-12-27): https://cdn.clinicaltrials.gov/large-docs/99/NCT04945499/Prot_000.pdf